CLINICAL TRIAL: NCT05182450
Title: Acute Effects of Mango Leaf Extract on Cognitive Function in Healthy Adults: A Double-Blind, Placebo-Controlled Crossover Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2102
Record Dates: First submitted 2021-11-16; First posted 2022-01-10 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Attention; Cognition; Mood
Keywords: mood; cognitive function; mango leaf; mango

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Capsules will disguise potential differences in colour/particle size of powders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active capsule (Experimental): Colored capsule containing 300 mg mango leaf extract (Zynamite®) standardized to contain ≥ 60% mangiferin. Supplied by PLT Health Solutions, Inc.
  Interventions: Other: Mango leaf extract capsule
- Placebo capsule (Placebo Comparator): Colored capsule, appearance-matched to the active experimental capsule
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Other: Mango leaf extract capsule — Single dose
  Arms: Active capsule
Other: Placebo capsule — Single dose
  Arms: Placebo capsule

SUMMARY:
The primary aim of this randomised, double-blind, placebo-controlled, cross-over study is to assess the short-term cognitive effects of a single dose (300 mg) of Mango Leaf Extract compared to a placebo on cognitive function, including during cognitively demanding task performance. The trial will utilise the COMPASS cognitive assessment system and cognitive demand battery (CDB), and Profile of Mood States (POMS), visual analogue mood scales (VAMS), and Stress Visual Analogue Scales (S-VAS) with assessments taking place at baseline, 30 minutes, 180 minutes and 300 minutes post treatment, on two separate testing days separated by 7 days (minimum).

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 45 years, inclusive
2. Self-reported good health
3. Willingness to abstain from consumption of caffeine within 12 h of testing
4. Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits
5. Willing to refrain from 'over the counter' medications (e.g., pain medication) and stimulant medication for 12 hours, seasonal allergy/hayfever nasal antihistamine medications for 24 hours and oral antihistamines for 48 hours prior to all test visits
6. Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator

Exclusion Criteria:

1. Failure to meet any one of the inclusion criteria
2. Have any pre-existing medical condition/illness which will impact taking part in the study, interact with the active treatments or impede performance
3. Current use of prescription medication (no antibiotics within the last 4 weeks) NOTE: the explicit exceptions to this are contraceptive treatments for female participants, and those taken 'as needed' in the treatment of asthma and hay fever. There may be other instances of medication use which, where no interaction with the active treatments is likely, and which would not be expected to have any impact on brain function, where participants may be able to progress to screening
4. Have sleep disorders or are taking sleep aid medication
5. Major trauma or major surgical event within 6 months of screening
6. Extreme dietary habits, as judged by the Investigator (high fat, very high protein diets, intermittent fasting, etc.)
7. Exposure to mango leaf extract (MLE) within 30 d prior to screening
8. History of cancer in the prior two years, except for non-melanoma skin cancer
9. Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour blindness)
10. Food allergies/intolerances/sensitivities to any ingredients in the study products and study meals (including related foods/beverages/products) and or unwillingness to eat or dislike for the study meals.
11. Self-report excessive leisure time physical activity (> 7 strenuous bouts per week)
12. Have a current or chronic gastrointestinal, sleep, or psychiatric disorders including medically diagnosed anxiety and depression
13. Work night shifts or follow a variable work pattern that results in irregular sleep pattern
14. Are pregnant, trying to get pregnant or lactating
15. Smoke tobacco, vape nicotine or use nicotine replacement products (including occasional social smoking)
16. Illegal/recreational drug use
17. Fail to demonstrate adequate minimal performance on lab, computer-based cognitive tasks
18. Have participated in another clinical trial within past 30 days and/or participation in another PepsiCo trial in the past 6 months
19. Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
20. Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2
21. Have a diagnosed neurological condition, or learning/behavioural or neurodevelopmental differences (e.g. dyslexia, autism, ADHD).
22. Excessive caffeine intake (>500 mg per day)
23. Have taken dietary supplements e.g. Vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4-week supplement washout prior to participating and for the duration of the study on the proviso that the supplements taken are out of choice and not medically prescribed or advised)
24. Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
25. Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
26. Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
27. Suffers from frequent migraines that require medication (more than or equal to 1 per month)
28. Any known active infections
29. Are non-compliant with regards treatment consumption
30. Does not have a bank account (required for payment)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of attention | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  Average % correct of attention tasks - choice reaction time, digit vigilance and 3 x rapid visual information processing task). Higher accuracy is better.

SECONDARY OUTCOMES:
General mood and psychological state, including depression and anxiety: VAMS | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  Visual Analogue Mood Scales (VAMS). Current subjective position marked on 100 mm lines anchored at either end by 18 antonyms (e.g. 'alert-inattentive', 'lethargic-energetic'). Better mood scores are a better outcome.
General mood and psychological state, including depression and anxiety: POMS | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  Profile of Mood States (POMS) consisting of 65 adjectives rated on a 0-4 scale. Better mood scores are a better outcome.
General mood and psychological state, including depression and anxiety: S-VAS | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  Stress Visual Analogue Mood Scales (S-VAS). Four items (anxious, stressed, relaxed, calm) rated not at all to extremely on 100 mm lines. Better mood scores are a better outcome.
Cognitive domain factor scores | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  Composite cognitive factors (speed of attention, working memory, speed of memory and episodic memory) averaged across individual tasks. Higher scores are better.
Global cognitive performance measures: Speed | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  Speed of cognitive performance comprising reaction time (msec) data averaged from all of the computerized cognitive assessment tasks that return speed data. Faster average speed is a better outcome.
Global cognitive performance measures: Accuracy | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  Accuracy of cognitive performance comprising % accuracy data averaged from all of the computerized cognitive assessment tasks that return accuracy data. Higher average % accuracy is a better outcome.
Cognitive performance: Episodic long term memory | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  A computerized series of individual cognitive tasks are presented on screen. Test components are word recall, word recognition and picture recognition. Better task performance is a better outcome.
Cognitive performance: Attention | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  A computerized series of individual cognitive tasks are presented on screen. Test components are choice reaction time, digit vigilance and simple reaction time. Better task performance is a better outcome.
Cognitive performance: Working memory | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  A computerized series of individual cognitive tasks are presented on screen. Test components are numeric working memory and corsi blocks. Better task performance is a better outcome.
Cognitive performance: Executive function | Change from pre-dose (baseline) to 30, 180 and 300 minutes post-treatment, comparing mango leaf to placebo
  A computerized peg and ball cognitive task is presented on screen. Better task performance is a better outcome.
Cognitive function and mental fatigue during extended performance of cognitively demanding tasks | 30, 180 and 300 minutes post-dose compared to placebo
  Cognitive Demand Battery (CDB) of component tasks: Serial 3s/7s, Rapid Visual Information Processing task (RVIP), Mental Fatigue Visual Analog Scale (VAS). 30 minute test (10 minute computerized assessment run three times in succession). Higher function and lower fatigue are better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Dodd, PhD, Principal Investigator — U. Northumbria, Brain Performance and Nutrition Research Centre, Department of Psychology
Locations (1):
- Northumbria University, Brain Performance and Nutrition Research Centre, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dodd FL, Kennedy DO, Johnson J, Haworth E, Greener JP, Jackson PA. Acute effects of mango leaf extract on cognitive function in healthy adults: a randomised, double-blind, placebo-controlled crossover study. Front Nutr. 2024 Apr 11;11:1298807. doi: 10.3389/fnut.2024.1298807. eCollection 2024. PMID 38665302